CLINICAL TRIAL: NCT02000986
Title: Effect of Non-Pharmacologic Interventions on Risk Factors of Cardiovascular Disease in Survivors of Childhood Leukemia, Lymphoma and Brain Tumor
Brief Title: Dietary and Exercise Interventions in Preventing Cardiovascular Disease in Younger Survivors of Leukemia, Lymphoma, or Brain Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-14062; HM14062 (Other: Virginia Commonwealth Unniversity IRB)
Record Dates: First submitted 2013-11-26; First posted 2013-12-04 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Childhood Brain Tumor; Childhood Hodgkin Lymphoma; Childhood Non-Hodgkin Lymphoma; Malignant Childhood Neoplasm
Keywords: Hodgkin's Lymphoma; Brain and Nervous System; Non-Hodgkin's Lymphoma; Leukemia, not otherwise specified
MeSH Terms: conditions — Neoplasms; Hodgkin Disease; Neurologic Manifestations; Lymphoma, Non-Hodgkin; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Specimen Collection/Risk Factor Assessment -> Diet/Exercise -> (Experimental): Specimen Collection/Risk Factor Assessment -> Diet/Exercise -> Chemotherapy
  Interventions: Behavioral: Specimen Collection/Risk Factor Assessment -> Diet/Exercise -> Chemotherapy

INTERVENTIONS:
Behavioral: Specimen Collection/Risk Factor Assessment -> Diet/Exercise -> Chemotherapy — Participants will be taught by a registered dietician about energy balance and how body weight relates to energy intake and expenditure, although specific calorie prescriptions will not be given. An exercise physiologist will create a personalized exercise plan and prescription which is tailored to his / her needs and current level of activity and fitness

SUMMARY:
This clinical trial studies dietary and exercise interventions in preventing cardiovascular disease in younger survivors of childhood cancer. Eating a healthy diet and exercising regularly may reduce the risk of cardiovascular disease in younger survivors of childhood cancer.

DETAILED DESCRIPTION:
Participants receive personalized exercise plan and prescription tailored to individual needs and current level of activity and fitness, and they also receive 2 one-hour individual exercise training sessions consisting of 20-30 minutes cardiovascular activity and strength training. Participants receive nutritional education consisting of energy balance, appropriate portion sizes, calorie count, and basic nutrition skills such as label reading every 2 weeks for 12 weeks.

After completion of study treatment, patients are followed for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pediatric cancer
* Patients 3 months to 1 year after completion of therapy

Exclusion Criteria:

* Patients who are already on antihypertensive or insulin or cholesterol lowering medication
* Patients who have not been evaluated for exercise tolerance and cleared by their physician for participation
* Inability to understand program instructions due to language barrier or mental disability
* Unable to participate in the outlined exercise program due to a physical disability

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Feasibility determined by average attendance and retention | At 3 months
  Acceptability will be determined by responses on feedback measures and qualitative analysis of exit interviews.

SECONDARY OUTCOMES:
Feasibility determined by average attendance and retention from the blood pressure at enrollment | At 6 months
  Will be assessed via paired T test.
Acceptability level at time of enrollment | At 6 months
  Acceptability will be determined by responses on feedback measures and qualitative analysis of exit interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Marieka A Helou, MD, Principal Investigator — Massey Cancer Center